CLINICAL TRIAL: NCT00450697
Title: Feeding Tolerance in Preterm Infants: Randomized Trial of Bolus Feeding Every 4 Hours Versus Every 3 Hours
Brief Title: Feeding Tolerance in Preterm Infants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Anita Stola, Weill Cornell MC
Other Study IDs: 0608008682
Record Dates: First submitted 2007-02-07; First posted 2007-03-22 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2010-11

CONDITIONS: Prematurity; Feeding Intolerance
Keywords: Feeding intolerance in premature infants; Bolus feeding every 4 hours versus every 3 hours; Feeding method in premature infants
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- observation

SUMMARY:
Premature infants, especially those less than 1250 gm at birth are extremely difficult to feed. For unknown physiologic reasons oral feeding also called enteral feeding is not well tolerated in these immature babies. Because of this challenge these infants require intravenous fluids solution called parenteral nutrition (TPN). Intravenous nutrition is inadequate because it cannot supply sufficient calories for growth both of body and brain. The composition of intravenous nutrition is also toxic to the liver.

For those reasons it is very important to achieve adequate enteral nutrition in premature infants as soon as possible after birth. However the best feeding method for those babies has not been defined.

Since premature babies are unable to suck and swallow properly, feeding is administered by a tube inserted into the infant's stomach. The timing between feeds is inconsistent. Some infants are fed every 3 hours, whereas others are fed every 4 hours.

The purpose of this study is to determine which feeding method is better. We hypothesize that feeding every 4 hours by allowing more time for digestion will improve feeding tolerance in premature infants. In addition it will also facilitate discontinuation of TPN sooner, thus causing less side effects.

DETAILED DESCRIPTION:
In premature infants feeding tolerance is limited due to immaturity of gastrointestinal tract. Motor patterns of the gastrointestinal tract differ greatly in preterm infants as compared to adults. These differences in gastrointestinal motor function in premature neonates translates into less efficient gastric emptying and slower intestinal transit time. It usually manifests as residual feeds in the stomach prior to the next scheduled feeding and may be associated with abdominal distention, bile-staining aspirates, or lack of stooling. In most instances the gastric residuals are benign and relate to immature gastrointestinal motility, however they may also be an early indication of bowel obstruction, ileus or necrotizing enterocolitis. Thus, feeding intolerance often leads to temporary cessation of feeds, and prolongs the time to reach full feeds, as well as the time on parenteral nutrition (which predisposes the infants to nosocomial infection, hepatic dysfunction), and prolonged hospitalization.

Achievement of adequate enteral nutrition, as soon as possible after birth is the ultimate goal for all low birth weight infants (<1250 gm); however the best methods by which sufficient enteral nutrition can be provided remain controversial.

A number of feeding strategies are practiced. In our Neonatal ICU feeds are initiated by boluses and infants are being fed either every 3 hours or every 4 hours. A review of the literature (2006) revealed that there was no study comparing those two methods of feeding. We hypothesize that very low birth weight infants (≤1250 gm) will tolerate feedings better when introduced every 4 hours instead every 3 hours, by providing sufficient time for gastric emptying.

We propose to conduct this prospective, randomized, clinical trial to determine whether intermittent bolus gavage feedings every 4 hours leads to better feeding tolerance than intermittent bolus gavage feedings every 3 hours in very low birth weight infants < 1250grams birth weight.

Primary Hypothesis:

Very low birth weight infants fed by intermittent bolus gavage every 4 hours will achieve full enteral feeding (120 kcal/kg per day) at an earlier postnatal age and have less feeding intolerance than infants fed every 3 hours.

Secondary Hypothesis:

Intermittent bolus gavage feeding every 4 hours will improve feeding tolerance, cause less need for parenteral nutrition and its major complication - cholestasis.

Study Design:

* Prospective, randomized clinical study with recruitment at NY Presbyterian Hospital Cornell Medical Center.
* Written informed consent will be obtained from one or both parents prior to enrollment of each patient.

Primary study endpoint:

* Days to reach full feeds of 120 ml/kg per day
* Incidence of feeding intolerance

Secondary study endpoint:

* Days on parenteral nutrition (parenteral nutrition is discontinued when an infant tolerates enteral feeding of 100 ml/kg per day).
* Incidence and severity of cholestatic jaundice.

Primary objective:

To determine whether infants fed by intermittent gastric bolus gavage every 4 hours will have less feeding intolerance and reach full feeds at least 2 days earlier than infants fed every 3 hours.

Secondary objectives:

To determine if feeding every 4 hours will facilitate discontinuation of parenteral nutrition at an earlier postnatal age and result in less incidence of cholestasis.

Inclusion Criteria Weight ≤ 1250 gm Sufficient stability to start early (day 3-5) enteral feedings Appropriate weight for gestational age Infants receiving ventilatory support and those with indwelling umbilical arterial catheters will be included Absence of major congenital malformations

Infant will be withdrawn from the study for the following reasons:

Parental request If feeding cannot be initiated prior to day of life 10 NEC requiring surgery Prolonged (> 3days) intolerance to the feeding regimen

Treatment plan:

Feeding Protocol

* Infants who meet all of the above criteria will be randomly assigned using sealed opaque envelopes, to either every the 3 hour or every 4 hour feeding groups.
* Nasogastric feeding will be initiated on the third to fifth postnatal day provided the infant's cardiorespiratory status is stable.
* Bolus feeding over 30 to 60 min will be given as per usual clinical practice
* Expressed breast milk is the nutrition of choice. If not available Premature Formula of 24 kcal/30 ml will be used as per usual clinical practice.
* Feeding will be started and advanced in daily increments depending on infant's weight:
* 500 gm to 750 gm - 10 ml/kg per day
* 751gm to 1000gm - 15 ml/kg per day
* 1001 gm to 1250gm - 20 ml/kg per day
* Gastric residual will be measured prefeed (every 3 or 4 hours)
* All feeding-related clinical decisions (when to withhold feedings) will be up to the attending physician's discretion.
* Parenteral nutrition, including lipid emulsion, will be started on days 1 or 2 and continued until each infant tolerates enteral feeding of 100 ml/kg per day.
* Successful achievement of full enteral feeding is defined as the ability to tolerate enteral feedings of 110-120 ml/kg per day for at least 48 hours.
* Daily weight, intake and output, number of stools, number of guaiac positive stools, number of hours that feedings were withheld, episodes of apnea and bradycardia will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Weight ≤ 1250 gm
* Sufficient stability to start early (day 3-5) enteral feedings
* Appropriate weight for gestational age
* Infants receiving ventilatory support and those with indwelling umbilical arterial catheters will be included
* Absence of major congenital malformations

Exclusion Criteria:

* Parental request
* If feeding cannot be initiated prior to day of life 10
* NEC requiring surgery
* Prolonged (> 3days) intolerance to the feeding regimen

Ages: 1 Day to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: very low birth weight premature infants with birth weight <= 1250g
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2007-02; Study Completion 2008-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Anita G Stola, MD, Principal Investigator — The New York Presbyterian Hospital-Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital; Weill Cornell Medical College; Department of Pediatrics; Division of Neonatology, New York, New York, United States